CLINICAL TRIAL: NCT01257295
Title: Properties of Dietary Fibre and Energy Intake: an Intervention to Study the Effect of Physicochemical Properties of Dietary Fibre on Energy Intake and Underlying Mechanisms
Brief Title: Properties of Dietary Fibre and Energy Intake
Acronym: ProVe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: METC-10/22
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2011-12-26 (Estimated); Status verified 2011-12

CONDITIONS: Healthy Male Subjects
Keywords: dietary fiber; energy intake; appetite; satiety hormones; glucose; gastric emptying
MeSH Terms: interventions — Breakfast

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- control (Placebo Comparator): No additions of fiber to a breakfast meal
  Interventions: Dietary Supplement: control: no fiber addition
- low viscous, low gelling (Active Comparator): low viscous, low gelling fibre added to breakfast meal
  Interventions: Dietary Supplement: breakfast with low viscous, low gelling pectin
- high viscous, low gelling (Active Comparator): high viscous, low gelling fibre added to breakfast meal
  Interventions: Dietary Supplement: high viscous, low gelling pectin
- low viscous, high gelling (Active Comparator): low viscous, high gelling fibre added to breakfast meal
  Interventions: Dietary Supplement: low viscous, high gelling pectin
- high viscous, high gelling (Active Comparator): high viscous, high gelling fibre added to breakfast meal
  Interventions: Dietary Supplement: high viscous, high gelling pectin
- fibre supplement (Active Comparator): high viscous, high gelling fibre is added, not to the breakfast meal, but as supplement
  Interventions: Dietary Supplement: pectin supplement

INTERVENTIONS:
Dietary Supplement: control: no fiber addition — liquid breakfast without addition of fiber
  Arms: control
Dietary Supplement: breakfast with low viscous, low gelling pectin — 10g of low viscous, low gelling pectin dissolved in a liquid breakfast
  Arms: low viscous, low gelling
Dietary Supplement: high viscous, low gelling pectin — 10g of high viscous, low gelling pectin dissolved in a liquid breakfast
  Arms: high viscous, low gelling
Dietary Supplement: low viscous, high gelling pectin — 10g of low viscous, high gelling pectin dissolved in a liquid breakfast
  Arms: low viscous, high gelling
Dietary Supplement: high viscous, high gelling pectin — 10g of high viscous, high gelling pectin dissolved in a liquid breakfast
  Arms: high viscous, high gelling
Dietary Supplement: pectin supplement — 10g of high viscous, high gelling pectin provided as a dietary supplement, a liquid breakfast is served seperately
  Arms: fibre supplement

SUMMARY:
Dietary fibers likely have a role in body weight management. They may increase satiety and, as a consequence, reduce energy intake during the next meal. There are, however, many different types of dietary fiber, which have diverse physical properties and can therefore impact these outcomes differently. It is, however, unclear whether dietary fibers with different properties lead to differences in energy intake during the next meal. The objective of this study is to study the effect of pectin in 4 different physicochemical states on ad libitum energy intake and possible underlying mechanisms; i.e. gastrointestinal hormones, gastric emptying rate, feelings of satiety and the method of fiber supplementation. We hypothesize that viscous and gelling fibers will reduce ad libitum energy intake compared to low viscous and low gelling fibers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30 year
* BMI 18.5-25 kg/m2
* Healthy as judged by the participant

Exclusion Criteria:

* Females
* Weight loss or weight gain of more than 5 kg during the last 2 months
* Using an energy restricted diet during the last 2 months
* Lack of appetite for any reason
* Restrained eater: >2.89, measured by DEBQ (35).
* Smoking
* Heavy alcohol use: >5 drinks/day (36).
* Reported stomach or bowel disease
* Reported diabetes
* Reported thyroid disease or any other endocrine disorder
* Reported intolerance for pectin, bread, gluten, dairy or not liking of the research foods
* Anemia: Hb<8.0 mmol/l
* Fasting glucose levels >5.8 mmol/l
* Blood donation from 6 weeks prior to the study until the end of the study
* Experienced any problems with drawing blood in the past
* Antecubital veins not considered suitable for blood drawing by means of a catheter
* Thesis students or employees of the division of Human Nutrition

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2010-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
energy intake | 3 hours
  3 hours after ingesting the test breakfast ad libitum energy intake is measured.

SECONDARY OUTCOMES:
appetite sensations | 3 hours
  appetite is measured by VAS scales over a period of 3 hours after ingestion of a test breakfast
satiety hormones | 3 hours
  satiety hormones (ghrelin, PYY, GLP-1, CCK) are measured over a period of 3 hours after ingestion of a test breakfast
gastric emptying rate | 3 hours
  gastric emptying rate is measured over a period of 3 hours after ingestion of a test breakfast
method of supplementation | 3 hours
  One of the fibers will be offered as tablets that will be ingested with a glass of water right after the test meal.

CONTACTS AND LOCATIONS:
Overall Officials: Edith Feskens, PHd, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Wageningen, Netherlands